CLINICAL TRIAL: NCT04154046
Title: Treatment of Impending Ulcers Associated With Hammer, Mallet and Claw Toe Deformities in the Diabetic Patient Setting
Acronym: TODDIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TODDIII
Record Dates: First submitted 2019-09-05; First posted 2019-11-06 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Foot; Hammer Toe; Mallet Toe; Claw Toe
MeSH Terms: conditions — Diabetic Foot; Hammer Toe Syndrome | interventions — Needles

STUDY DESIGN:
Intervention Model Description: Patients WHO meet all inclusion and non of the exclusion criteria are randomly allocated to two arms in the study. The allocation is stratified by treatment center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenotomy (Experimental): Patients allocated to this arm receive tenotomy treatment of affected toes, and standard care including offloading treatment
  Interventions: Procedure: Tenotomy(cutting) of flexor tendons is performed with needle
- standard care (No Intervention): Patient who are randomized to this arm receive standard care including offloading treatment

INTERVENTIONS:
Procedure: Tenotomy(cutting) of flexor tendons is performed with needle — Patient is placed in seated posture with feet elevated. The toe(s) with hammer, mallet or claw toe deformity is anesthetized by a digital toe block with 1-5 ml of 1% lidocaine administered for each toe. The toe digital block is administered through a plantar approach, at the web level of the deformed toe(s), with a 0,6 mm diameter and 30mm long needle.
  After anesthetizing the toe(s) the plantar aspect of the toe at web level is disinfected with an alcohol based disinfectant twice.
  Both the long and short flexors are then severed with a 1.2mm diameter and 40mm long needle through a plantar approach, immediately proximal to the web level of the toe.
  After the procedure a dry gauze bandage is applied and the patients treated foot/feet is/are elevated for 20 minutes to achieve haemostasis, and the bandage is checked for bleeding before discharge.
  Arms: Tenotomy

SUMMARY:
Patients with diabetes, hammer, mallet and claw toes and impending ulcers associated with hammer mallet and claw toes will be randomized to tenotomy (cutting) of flexor tendons to the afflicted toes, done by needle and standard offloading or offloading alone. Impending ulcers are defined as callus or nail changes that are known pre-stages to ulcers. The effects of the surgery on incidence of ulcers associated with the named deformities, and rate of complications associated with the surgery.

DETAILED DESCRIPTION:
1. STUDY RATIONAL Diabetes is one of the largest medical challenges facing the world today. 12% of the world's health budget is spent on diabetes, that is USD 673 billion (Euros 585 billion). It is estimated that a lower limb is amputated due to diabetes every 30 sec. on a global scale, and it is known that 85% of all amputations are performed due to a diabetic ulcer1. In Denmark 320.000 citizens has a diabetes diagnosis, an additional 200.000 are estimated to have diabetes unknowingly, and 750.000 to have the pre-stages of diabetes2. These numbers have doubled in the past ten years and are estimated to cost DKK 86 million a day (or Euros 11.6 million a day)1. One of the complications to diabetes is the "diabetic foot syndrome", which is a result of neurological abnormalities, vascular complications or a combination of the two. Knowledge about the causes of the disease has been gathered since the late nineteenth century3. In recent years, preventive therapy has been the focus of treatment, resulting in several national and international guidelines4,5,6. Focus has been on education in self-care and awareness of risk factors, combined with "Foot-at-Risk" evaluation7, at least once a year and off-loading therapy crafted and applied by specialized personnel3,4.

   Steno Diabetes Center Copenhagen, University of Copenhagen, Denmark is a highly-specialized treatment facility focusing on the patient with diabetes. In spite of optimized treatment for patients with diabetes, and the fact that incidence of first time ulcers in patients with type 1 and 2 diabetes is declining, the incidence of first time ulcers is still 2.6 and 8.7 per. 1000 patient years for type 1 and 2, respectively8. Diabetic foot ulcers have a known association with increased mortality, morbidity and economic burden9,10,11, at the same time most amputations in patients with diabetes are preceded by an ulcer12.

   Hammer, mallet and claw-toe deformities are some of the most common deformities associated with the diabetic foot syndrome. Prevalence has been reported between 32% and 46%13,14. These deformities are predictors of diabetic foot ulcers15,16. There are several theories on the etiology of hammer, mallet and claw toe deformities - the three classic deformities of the toes. In the diabetic patient setting, the classical theory is based on neuropathy (nerve damage associated with diabetes and other diseases), resulting in intrinsic muscle (muscles of the foot) dysfunction, changes that lead to imbalance between the flexor and extensor tendons, which in turn leads to hyperextension of the metatarsophalangeal (MTP) joint and/or flexion in the interphalangeal joints (IP), leading to the three classic deformities of the toes. The neuropathic theory is not sufficient to explain the full scope of the problem 4, and other theories have been proposed17. In the non-diabetic patient, the neuropathic explanation is not viable, but the explanations still center on an imbalance between in- and extrinsic musculature, resulting from deformities in the foot either as flexor-substitution or stabilization deformities18. The deformities change the pressure on the plantar aspect of the foot19. These changes in pressure make specific contact points predilection sites for ulcers. The sites have been described as tip of the toe ulcers, cock-up ulcers, kissing ulcers and plantar metatarsal ulcers20.

   The treatment of hammer, mallet and claw toe deformities in diabetes has classically consisted of offloading in the form of shoes, insoles and/or orthosis (i.e. silicone spacers, felt pads etc.) or flexor tendon tenotomy (cutting tendons) done by scalpel. Several studies on flexor tenotomies performed with scalpel have been performed21,22; all have reported acceptable or positive results on ulcer healing and low complication rates, including one study from our own institute23. At Diabetic Foot Study Group 2018 we presented unpublished results from a study showing that tenotomy done by needle has comparable results to the classical scalpel. However, no study has, to our knowledge, been published comparing conservative treatment with surgical approach to these deformities, let alone randomized controlled trials (RCT).
2. WHAT DOES THIS TRIAL ADD TO CURRENT KNOWLEDGE? This is to our knowledge the first RCT looking at flexor tenotomies as a preventive treatment, and/or compared to conservative treatment. At the same time this is the first study looking at needle flexor tenotomies, as opposed to the classic tenotomies done by scalpel.
3. HYPOTHESIS We hypothesize that treating hammer, mallet and claw toe deformities in patients with type 1 and 2 diabetes, and impending ulcers (defined as nail changes, and hypercallosities at the predilection sites for ulcers associated with hammer, mallet and claw toe deformities) with needle tenotomy is a safe and effective treatment, and superior compared to offloading (conservative) treatment done by silicon spacer, insoles, felt, and/or therapeutic sandals
4. AIM The aim of the RCT is to evaluate the effect of needle tenotomy when treating impending ulcers associated with hammer, mallet and claw toe deformities.

   The study is designed as a prospective RCT comparing needle tenotomy with conservative treatment, for patients with deformities and impending ulcers associated with the three deformities.

   Primary endpoint will be number of new ulcers incurred, defined as ulcers associated with hammer, mallet and claw toe deformities, placed on treated foot.

   Secondary endpoints will be complications: infections (defined as ailment associated with procedure or ulcer, that is diagnosed as infection by attending health professional), transfer lesions (defined as impending ulcers or actual ulcers at anatomical sites associated with hammer, mallet and claw toes in patients with diabetes, on non-treated hammer, mallet and claw toes after surgical treatment), minor amputations (defined as amputations below ankle level), major amputations (defined as amputations at or above ankle level).
5. STUDY I 5.1 Design A prospective RCT involving patients with diabetes as well as one of the three deformities and an impending ulcer associated with the mentioned deformities. By randomization, patients will be allocated to either conservative treatment or tenotomy performed by needle.

   5.2 Statistical analysis plan Sample-size The calculation is done with a Type 1 error rate at 5%, and a power at 80%. The primary endpoint is number of new ulcers incurred.

   In the general diabetic population life time prevalence of diabetic ulcers has been reported at 15-25%24, the yearly incidence in the same group is 6%. This study focuses on patients with a deformity reported to have a 1.5 hazard ratio25, and signs of an impending ulcer like callus formation, which has been reported with a relative risk of 1126. The incidence of new diabetic foot ulcers incurred by the study population is set at 10%, according to the above mentioned considerations.

   The incidence in the intervention group is set at 6%, so the anticipated reduction in incidence is 4% compared to the incidence in the control group which as above mentioned is set at 10%.

   However, the numbers for incidence of new diabetic foot ulcers is an uncertain size, especially when looking at the specific group we are looking at, therefore the standard deviation is set at 10.

   The calculator used is a 2 means, 2 sample, 2-sided equality calculator. The formula is 18 With the above described parameters, the sample size is 98 patients, which due to an expected dropout of 10% will be extended to 110 patients.
6. PERSPECTIVE The results of these studies will allow us to evaluate if there's a clinical advantage to performing preventive tenotomies. Several studies have shown that tenotomies done by scalpel are safe, and that most patients go on to heal their ulcers, but none have compared tenotomies to standard care, and no studies have looked at tenotomies as a preventive treatment against new ulcers. Our hypothesis is that patients with impending ulcers associated with hammer, mallet and claw toe deformities will have a lower incidence of new ulcers associated with hammer, mallet and claw toe deformities. At the same time, unpublished data from our institute show that tenotomies done by needle has comparable results to tenotomies done by scalpel. The economic perspectives are vast if a preventive minimal invasive procedure, that can be performed in everyday clinical work, with a minimal surgical technique requirement, can lead to significant reductions in incidence of new ulcers.
7. QUALITY CONTROL AND MONITORING The studies will be performed in accordance with the Helsinki Declaration, International Council for Harmonization of technical requirements for pharmaceuticals for human use (ICH) Guidelines for good Clinical Practice (GCP)27. and after approval by the The National Committee on Health Research Ethics and the Data Monitoring Board in Denmark. The study will be registered on http://www.clinicaltrials.gov/.

   Permission for a third person to have access to patient data will be obtained at screening visit. Investigators will provide access to source data and relevant documents in connection with monitoring, inspections, and audits to all relevant authorities.
8. ETHICAL CONSIDERATIONS AND DATA SAFETY The study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki 1996 and the principles of GCP28 8.1 Ethical committee approval The appropriate approval from a local Danish ethical committee will be obtained before start of trial, and their guidelines will be followed throughout the process. Patients will receive oral and written information on the study, before being required to sign an informed consent paper.

   8.2 Personal data usage and protection The appropriate approval from the Danish data protection agency will be obtained before the study commences, and their guidelines will be followed throughout the process. All patient data will be stored and treated in accordance with regulation 2016/679 from the European parliament on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, dated 27 April 201629, and the Danish amendment to regulation 2016/67930.

   8.3 Patient Perspective Patients enrolled in this study will receive a treatment that is already implemented in our and several other clinics, and the unpublished data from our retrospective study and the formerly published data on tenotomies, points towards tenotomies being a safe and effective treatment of hammer, mallet and claw toes. Patients who don't receive intervention in the form of tenotomies in the study, will receive standard offloading and ulcer treatment, and be offered to undergo tenotomy if an ulcer occurs and tenotomi is found relevant. In conclusion the patients enrolled in the study will receive a treatment with potential benefits for them, and a low risk of complications making the study ethically sound.
9. RECRUITMENT Patients will be recruited and treated at the three study sites, Bispebjerg Hospital, Hilleroed Hospital and Steno Diabetes Center Copenhagen. Healthcare professionals (doctors, nurses and podiatrists) with daily care of patients with diabetes will be encouraged to look for potential study candidates in the outpatient clinics. If any potential candidates are found, patients will receive written information on the project, asked if we can contact them regarding the study and referred to one of the investigators for further screening. When referred to investigator, eligibility criteria will be confirmed based on information from the patients' electronic record (sundhedsplatformen). Patients will hereafter be contacted by telephone. If patients do not respond to contact by telephone, they will be contacted by letter.

   In addition to the above mentioned method, primary investigator will conduct a screening of patients that are currently treated at the three institutes for eligible candidates. This screening will be conducted through the patient electronic record (sundhedsplatformen). The data that is screened in patient electronic record, includes all data relevant for in/exclusion criteria, namely prior diagnosis, operations, medicine use and visit information.

   Identified candidates will be contacted by letter. If patients do not respond to letter, they will be contacted by phone.

   Before written consent is given, patients will be informed orally and in writing by the educated study personnel, including information on procedures, visits, goal of the study, and their rights as participants.

   General practitioners will be contacted by mail and asked to refer likely candidates to relevant study site (i.e. Hilleroed, Bispebjerg or Steno). The general practitioners and licensed podiatrists in the region will be informed by standard text, in the form of a standard letter To increase potential candidates found, adds in relevant locale newspaper and in national magazines. The ads will be in standard texts.

   Written consent will be acquired at inclusion visit by study related personnel. Patients will be required to fill out written consent form, after they have received oral and written information and been allowed up to 24 hours consideration and the possibility of bringing a personal assessor to participate at information and screening visits. If the patient needs additional time to consider, a follow-up meeting will be arranged minimum 24 hours after the first visit. Patients are informed that they can always withdraw their commitment to participate in the study, without consequences for their further treatment. No study related procedures are done until informed consent is signed by the patient.
10. DISSEMINATION OF RESULTS The study is initiated by Peter Rossing. Data is owned by the investigators. Positive, inconclusive as well as negative study results will be published in both national and international oral and written presentations as well as peer-reviewed international scientific journals. If data against expectations are not published in international journals, positive as well as negative study results will be published on a public website, for example www.clinicaltrials.gov.
11. PATIENT INFORMATION

11.1 Written Information All patients will receive information detailing the project, written information on their rights as Participants in research projects from the Danish ethics committee31, and written information on the procedure, potential unintended side effects, and what to expect after the operation.

11.2 Verbal Information All patients will be informed in layman's terms on the details of the operations, potential unintended side effects, and what to expect after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Type 1 or 2 diabetes
* Hammer, mallet or claw toe deformity
* Impending ulcer associated with above mentioned deformities
* Able to understand written and oral information
* Ability to follow planned visits and treatment
* Able to provide informed consent in Danish and/or English

Exclusion Criteria:

* Revascularization procedure in the affected limb planned, or undertaken within the 4 weeks prior to screening
* Hammer, mallet and claw toe that are rigid in both MTP and IP joints
* Ulcer associated with hammer, mallet and claw toe deformities
* Toe pressure < 30mmHg
* Prior major amputations on affected or ipsilateral leg
* Other corrective operation is indicated to treat patients foot deformities as deemed by investigator
* Current treatment with cytotoxic drugs or with systemically administered glucocorticoids
* Treatment of foot ulcers with growth factors, stem cells or equivalent preparations within the 8 weeks prior to screening
* Likely inability to comply with the need for planned visits because of planned activity
* Participation in another interventional clinical foot ulcer-healing trial within the 4 weeks prior to screening
* Prior enrolment in this trial
* Judgement by the investigator that the patient does not have the capacity to understand the study procedures or provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
New ulcers incurred | 1 year
  Number of new ulcers incurred, defined as ulcers associated with hammer, mallet and claw toe deformities, placed on treated foot

SECONDARY OUTCOMES:
Incidence of minor amputations | 1 year
  Incidence of minor amputations
Incidence of major amputations | 1 year
  Incidence of major amputations
incidence of secondary infection | 1 year
  incidence of secondary infection as deemed by treating physician
Transfer lesion incidence | 1 year
  Transfer lesions defined as impending ulcers or actual ulcers at anatomical sites associated with hammer, mallet and claw toes in patients with diabetes, on non-treated hammer, mallet and claw toes after surgical treatment)
Incidence of new ulcers on feet | 1 year
  Measured in incidence of new ulcers, defined as ulcer in different anatomical position than the treated ulcer(s) and associated with hammer, mallet or claw toes

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Hospitalerne i Nordsjælland Hillerød Hospital Ortopædkirurgisk afdeling, Hillerød
  - Videncenter for Sårheling Bispebjerg Hospital, København NV

IPD SHARING:
Plan to Share IPD: Yes
Protocol, ICF, and SAP will be shared when possible
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol, SAP and ICF shared here

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT04154046/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT04154046/ICF_000.pdf